CLINICAL TRIAL: NCT00003953
Title: A Phase II Study of Preoperative Dose-Dense Chemotherapy With Sequential Doxorubicin and Docetaxel for Initial Treatment of Operable and Inoperable Stage II-IIIB Breast Cancer
Brief Title: Chemotherapy Followed by Surgery in Treating Women With Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU2198; P30CA043703 (NIH); CWRU-2198 (Other: Case Comprehensive Cancer Center); NCI-G99-1537
Record Dates: First submitted 1999-11-01; First posted 2004-04-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; CMF regimen; Cyclophosphamide; Methotrexate; Fluorouracil; Docetaxel; Doxorubicin; Tamoxifen; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxorubicin and Docetaxel (Experimental)
  Interventions: Biological: filgrastim; Drug: CMF regimen; Drug: docetaxel; Drug: doxorubicin hydrochloride; Drug: tamoxifen citrate; Procedure: autologous bone marrow transplantation; Procedure: surgical procedure; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Filgrastim (G-CSF) is administered subcutaneously on days 3-10 of each 2 week course.
Drug: CMF regimen — Stratum I and II: receive cyclophosphamide, methotrexate, and fluorouracil (CMF) for 4 courses
  Other Names: cyclophosphamide; methotrexate; fluorouracil
Drug: docetaxel — Docetaxel IV over 1 hour on days 43, 57, and 71.
Drug: doxorubicin hydrochloride — Doxorubicin IV on days 1, 15, and 29.
Drug: tamoxifen citrate — Patients with positive estrogen or progesterone receptors receive oral tamoxifen daily for 5 years.
Procedure: autologous bone marrow transplantation — Stratum III:may receive high dose chemotherapy with stem cell support
Procedure: surgical procedure — Fourteen to 21 days following preoperative chemotherapy, patients undergo a radical, modified radical, or breast sparing surgery plus axillary lymph node dissection.
Radiation: radiation therapy — Radiotherapy is administered 5 days a week for 5.5 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of doxorubicin and docetaxel followed by surgery in treating women who have stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical and pathological response of women with stage II-IIIB primary breast cancer to preoperative high dose chemotherapy with sequential doxorubicin and docetaxel. II. Determine the safety and toxicity of this regimen in these patients. III. Determine the rate of breast conservation surgery in these patients on this regimen. IV. Determine the clinical response of these patients to docetaxel after 3 courses of doxorubicin. V. Correlate any circulating tumor cells shed at time of surgery with clinical response and pathological findings in these patients. VI. Determine whether tumor response correlates with HER2/neu expression of the primary tumor.

OUTLINE: Patients receive doxorubicin IV on days 1, 15, and 29, followed by docetaxel IV over 1 hour on days 43, 57, and 71. Filgrastim (G-CSF) is administered subcutaneously on days 3-10 of each 2 week course. Fourteen to 21 days following preoperative chemotherapy, patients undergo a radical, modified radical, or breast sparing surgery plus axillary lymph node dissection. Patients with disease progression or inoperable stage IIIB disease are removed from study. Following surgery, patients are stratified into one of three postoperative regimens: Stratum I: Patients with 0 lymph node metastases receive no further chemotherapy or receive cyclophosphamide, methotrexate, and fluorouracil (CMF) for 4 courses. Stratum II: Patients with 1-3 lymph node metastases receive CMF for 4 courses. Stratum III: Patients with at least 4 lymph node metastases or stage IIIB may receive high dose chemotherapy with stem cell support. Two to 6 weeks after surgery, patients undergoing breast sparing procedure receive adjuvant radiotherapy. Patients undergoing mastectomy receive chest wall and supraclavicular radiotherapy if initial clinical stage is T3, T4, or N2. All other patients with N1 with greater than 4 lymph nodes and N3 should receive radiotherapy. Radiotherapy is administered 5 days a week for 5.5 weeks. Patients with positive estrogen or progesterone receptors receive oral tamoxifen daily for 5 years. Patients are followed every 3 months for 3 years, then every 6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 27-35 patients will be accrued for this study.

ELIGIBILITY:
Eligibility Criteria:

* Women with a diagnosis of breast cancer established by tissue obtained by needle biopsy or incisional biopsy.
* There must be a residual measurable breast and/or axillary mass after biopsy.
* Clinical stage T1, N1-3, Mo or T2-4, N0-3, Mo. T2N0 lesions < 4cm in maximum dimension are eligible only if breast conservation is not feasible or practical without preoperative tumor shrinkage.
* Patients must be willing to undergo a mastectomy or breast sparing procedure plus axillary lymph node dissection.
* There must be no evidence of systemic metastases.
* No prior chemotherapy. Patients may have received up to 14 days of tamoxifen. 3.1.7 Patients > 18years are eligible.
* ECOG performance status 0-1.
* Normal hematologic function defined as white blood cell count > 3500/111 or neutrophil count > 1500411 and platelets >100,000/4
* Normal renal function defined as serum creatinine <1.5 mg/di.
* Adequate hepatic function. Bilirubin must be < institutional upper limit of normal (ULN). Transaminases (SGOT and/or SGPT) may be up to 2.5 X institutional ULN if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 4 X ULN if transaminases are < ULN. However, patients who have both transaminase elevation > 1.5 X ULN and alkaline phosphatase > 2.5 X ULN are not eligible for this study (due to decreased clearance of docetaxel and increased risk of toxicity).
* Patients with prior CIS of cervix or nonmelanoma skin cancers are eligible. Patients with prior DCIS or LCIS of breast are eligible if not previously treated with radiation or chemotherapy. Patients with prior malignancies including contralateral breast cancers treated with curative intent more than 5 years before enrollment are eligible.
* Patients must have signed informed consent.

Exclusion Criteria:

* Patients with a prior history of malignancy other than those mentioned in section 3.1.12 are ineligible.
* Patients must not have severe concurrent medical or psychiatric illness (i.e. no severe diabetes mellitus, poorly controlled ischemic heart disease or congestive heart failure, or severe chronic obstructive or restrictive pulmonary disease).
* The interval between initial diagnosis of breast cancer and the start of treatment must not be greater than 8 weeks.
* Due to anticipated toxicities to an unborn fetus, and excretion of chemotherapy in breast milk, patients must not be pregnant or lactating and must use effective contraception during treatment.
* No history of hypersensitivity reaction to preparation containing polysorbate 80, 3.2.6 Patients must not have peripheral neuropathy grade 2 or higher.
* Patients must not have had prior radiation to >25% of bone marrow

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1999-02; Primary Completion 2001-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determine the clinical response of these patients to treatment | after 3 courses (12 weeks)
  A clinical evaluation of tumor size includes repeat measurements of the palpable tumor in 2 dimensions, repeat mammography, if originally informative, of the affected breast with measurements of the palpable tumor in 2 or 3 dimensions and/or, evaluation of ipsilateral axillary lymph nodes with measurements, if palpable.
Pathological Response | after surgery at 15 weeks
  Number of patients with a complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD). CR is defined as disappearance of lesions. PR is defined as at least a 50% reduction in the sum of lesions. SD is defined as no significant change and PD is defined as the increase in the size of lesions.

SECONDARY OUTCOMES:
Detection of circulating tumor cells | after surgery at 15 weeks
  Detection of circulating tumor cells will be done using a panel of immunocytochemical antibodies directed against breast cancer epithelial cells and IMPATH/BIS laboratories. This assay can detect as few as 1 in 5x105 circulating tumor cells
Tumor response correlates with HER2/neu expression of the primary tumor. | baseline
  Pretreatment core needle biopsies will be analyzed for expression of HER2/neu expression using immunohistochemical staining.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda W. Cooper, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Metro Health Medical Center, Cleveland, Ohio

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=cwru2198